CLINICAL TRIAL: NCT04069949
Title: An Exploratory Study of Sorafenib Plus Toripalimab for Unresectable Hepatocellular Carcinoma With Portal Vein Tumor Thrombus
Brief Title: Sorafenib Plus Toripalimab for Unresectable HCC With Portal Vein Tumor Thrombus
Acronym: STUHCCPVTT
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Zhen-Yu Ding, Professor, Sichuan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LQ108
Record Dates: First submitted 2019-08-24; First posted 2019-08-28 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Unresectable Hepatocellular Cancer; Portal Vein Tumor Thrombus
Keywords: Sorafenib; Toripalimab; Unresectable; Hepatocellular Cancer; Portal Vein Tumor Thrombus
MeSH Terms: conditions — Liver Neoplasms | interventions — Sorafenib; toripalimab

STUDY DESIGN:
Intervention Model Description: one-arm study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- sorafenib plus toripalimab (Experimental): Stage I：Subjects (n=3) in cohort A received oral sorafenib (400 mg qd), in combination with intravenous toripalimab (240 mg d1, q3w). Subjects (n=3) in cohort B received oral sorafenib (400 mg bid) and the administration of toripalimab is consistent with cohort A. If dose-limiting toxicity (DLT) does not occur within 42 days of the first administration, the dose is escalated.
  Stage II: According to the expansion dose based on stage I, subjects are enlarged to 39.
  Interventions: Drug: sorafenib; toripalimab

INTERVENTIONS:
Drug: sorafenib; toripalimab — Stage I: cohort A: sorafenib 400 mg qd+ toripalimab 240 mg d1; q3w cohort B: sorafenib 400 mg bid, toripalimab 240 mg d1; q3w Stage II: According to the expansion dose based on stage I, subjects are enlarged to 39.

SUMMARY:
This study aims to evaluate the efficacy and safety of sorafenib plus toripalimab for unresectable hepatocellular carcinoma (HCC) with portal vein tumor thrombus (PVTT).

DETAILED DESCRIPTION:
Investigators aimed to conduct an exploratory study- an open-label, single-arm and multi-center -to evaluate the efficacy and safety of sorafenib plus toripalimab for unresectable hepatocellular carcinoma (HCC) with portal vein tumor thrombus (PVTT). The primary objectives are 6-month progression free survival (PFS) rate and safety. Secondary objectives include objective response rate (ORR), disease control rate (DCR), progression free survival (PFS), overall survival (OS) and duration of response. The study is divided into dose escalation stage and expansion stage.

Stage I (escalation stage) was designed to identify the dose-limiting toxicity (DLT) of the combination therapy. Subjects enrolled were divided into two cohorts. Subjects (n=3) in cohort A received oral sorafenib at doses of 400 mg once daily, in combination with intravenous toripalimab 240 mg on the first day, every 3 weeks. Subjects (n=3) in cohort B received oral sorafenib at doses of 400 mg twice daily, in combination with intravenous toripalimab 240 mg on the first day, every 3 weeks. If DLT does not occur within 42 days of the first administration, the dose is escalated. If one subject experienced DLTs, additional 3 subjects are enrolled at that level. Unless no DLT occurs, the next dose level test is continued.

Once ≥2 subjects in cohort A experienced DLT, the study is suspended in advance. If ≥2 subjects in cohort B experienced DLT, the dose of cohort A is recommended in expansion stage. If DLT does not occur in cohort B or only 1 of 6 subjects suffered DLT, the dose of cohort B is recommended in expansion stage.

For subjects who experienced DLT, if adverse events (AEs) return to normal or common terminology criteria for adverse events (CTCAE) level 1 within 2 weeks and researchers believe continuing treatment is beneficial to the subjects, they can continue treatment after dose adjustment. Otherwise, termination of treatment is suggested.

According to CTCAE version 4.0, DLT was defined as any grade ≥3 treatment-related toxicity occurring within the first 42 days of administration. Six to twelve patients will be included in this stage.

Stage II (Expansion stage): According to the expansion dose based on stage I, subjects are enlarged to 39. Subjects enrolled are treated with oral sorafenib in combination with toripalimab (every 3 weeks) until suffering progressive disease (PD) or un-tolerated toxicities. Previous literature indicated 6-month PFS rate for HCC with PVTT treated with sorafenib is about 20%. Investigators hypothesize sorafenib plus toripalimab could improve 6-month PFS rate to 40%. Software (PASS) is used to calculate the sample size (β=0.2，α=0.05). According to the results, 35 subjects should be enrolled. When 10% missing rate is considered, total subjects is 39.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic or cytologic diagnosis of unresectable hepatocellular carcinoma, or confirmed clinically in accordance with Chinese Association for the Study of Liver Diseases criteria (v2017)
2. Radiographically measurable disease by RECIST version 1.1 in at least one site
3. Radiographic evidence of portal vein cancer thrombus
4. Survival expectation ≥3 months
5. Eastern Cooperative Oncology Group: 0 or 1
6. Child-Pugh score A or B: score ≤7
7. Not previously treated with any systemic anti-cancer treatment (i.e. chemotherapy, target drugs, immune checkpoint inhibitors); Subjects who have received local hepatic therapy such as surgery, ablation, radiotherapy or transcatheter arterial chemoembolization, progression of target lesions after local treatment is required to increase by 25%, or target lesions are untreated, and the end of local treatment is more than 4 weeks.
8. All eligible patients have adequate organ function (ANC ≥1.5× 10⁹ / L, PLT ≥75 × 10⁹ /L, HGB≥90 g/L (no blood transfusion or EPO tolerance within 7 days), Cr≤1.5 times the ULN, TBN ≤1.5 times ULN, ALT and AST ≤3 times ULN, albumin ≥30g/L (albumin or branched chain amino acids supplementation is not allowed within 14 days), INR≤1.5 times the ULN, Urine protein≤1+).
9. Signed and dated written informed consent

Exclusion Criteria:

1. History of severe allergic reactions to chimeric, human or humanized antibodies, or fusion proteins. Hypersensitive to any component of the CHO cell-derived preparation or JS001 preparation
2. Pregnant or lactating women, men and women of childbearing age who are unwilling or unable to take effective contraceptive measures
3. History of other malignancy within the past 5 years
4. Medium or more pleural and ascites with clinical symptoms
5. Active hemorrhage or abnormal coagulation function (PT>16s, APTT>43s, INR>1.5 x ULN), or having a tendency to bleed or undergoing thrombolysis, anticoagulation or anti-platelet therapy
6. Central nervous system metastases
7. Hepatic encephalopathy
8. History of gastrointestinal bleeding or having a tendency to bleed within 6 months before enrollment, e.g. local active ulcer lesions; fecal occult blood (+ +) or above should not be included; if continuous fecal occult blood (+), gastroscopy should be performed.
9. Gastric or esophageal varices requiring treatment
10. Untreated active hepatitis B (i.e. subjects with hepatitis B undergoing antiviral therapy and HBV Load < 100IU/mL before the first administration of Toripalimab , is allowed to be enrolled; for subjects with anti-HBc (+), HBsAg (-), anti-HBs (-) and HBV viral load (-) , prophylactic anti-HBV therapy is not required, but virus activation should be closely monitored)
11. HCV and the anti-HCV treatment ended within 4 weeks of the first administration. Notably, subjects with untreated chronic HCV infection or untreated HCV are allowed.
12. History of drug abuse or mental disorders
13. History of organ or marrow transplants, or active autoimmune diseases requiring systemic treatment occurred within 2 years of the first administration
14. Immunodeficiency disorders or HIV
15. Pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonia, drug-related pneumonia and severe impairment of pulmonary function
16. Using immunosuppressive agents or systemic or absorbable local corticosteroids for immunosuppressive purposes (prednisone or its equivalent at dose> 10 mg/day) , and the above are used within 2 weeks before admission.
17. Major liver or other operations were performed within 4 weeks of the first administration, or minor operations were performed within 1 week before the first administration (simple excision, tooth extraction, etc.)
18. Receiving vaccine within 30 days of the first administration
19. Abdominal fistula, gastrointestinal perforation or abdominal abscess within 4 weeks of the first administration
20. Receiving other experimental drugs or medical devices within 4 weeks of the first administration
21. Any significant clinical and laboratory abnormalities that in the opinion of the investigator would affect safety assessment
22. Failure to satisfy the investigator of fitness to participate for any other reason.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
6-month Progression Free Survival rate | up to 6 months
  Proportion of patients with Progression Free Survival in 6-month
Incidence of Treatment-Emergent Adverse Event | up to 6 months
  Any adverse events related with treatment with Sorafenib Plus Toripalimab

SECONDARY OUTCOMES:
Objective Response Rate | up to 6 months
  Proportion of patients whose tumor volume has reached a predetermined value and can maintain a minimum time limit, including complete response and partial response patients
Disease Control Rate | up to 6 months
  Proportion of patients with stable disease, complete response and partial response
Progression Free Survival | up to 6 months
  A duration from the date of initial treatment with Sorafenib Plus Toripalimab to disease progression (defined by RECIST 1.1) or death of any cause.
Overall Survival | up to 1 year
  Duration from the date of initial treatment with Sorafenib Plus Toripalimab to the date of death due to any cause.
Duration of response | From the date of study enrollment to the time of death from any cause, assessed up to 1 year
  time from first documented complete or partial response to radiologically confirmed disease progression or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Qiu Li, Professor, Principal Investigator — West China Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Torre LA, Bray F, Siegel RL, Ferlay J, Lortet-Tieulent J, Jemal A. Global cancer statistics, 2012. CA Cancer J Clin. 2015 Mar;65(2):87-108. doi: 10.3322/caac.21262. Epub 2015 Feb 4. PMID 25651787
- [Background] Zhang ZM, Lai EC, Zhang C, Yu HW, Liu Z, Wan BJ, Liu LM, Tian ZH, Deng H, Sun QH, Chen XP. The strategies for treating primary hepatocellular carcinoma with portal vein tumor thrombus. Int J Surg. 2015 Aug;20:8-16. doi: 10.1016/j.ijsu.2015.05.009. Epub 2015 May 27. PMID 26026424
- [Background] Schoniger-Hekele M, Muller C, Kutilek M, Oesterreicher C, Ferenci P, Gangl A. Hepatocellular carcinoma in Central Europe: prognostic features and survival. Gut. 2001 Jan;48(1):103-9. doi: 10.1136/gut.48.1.103. PMID 11115830
- [Background] Pawarode A, Voravud N, Sriuranpong V, Kullavanijaya P, Patt YZ. Natural history of untreated primary hepatocellular carcinoma: a retrospective study of 157 patients. Am J Clin Oncol. 1998 Aug;21(4):386-91. doi: 10.1097/00000421-199808000-00014. PMID 9708639
- [Background] Llovet JM, Ricci S, Mazzaferro V, Hilgard P, Gane E, Blanc JF, de Oliveira AC, Santoro A, Raoul JL, Forner A, Schwartz M, Porta C, Zeuzem S, Bolondi L, Greten TF, Galle PR, Seitz JF, Borbath I, Haussinger D, Giannaris T, Shan M, Moscovici M, Voliotis D, Bruix J; SHARP Investigators Study Group. Sorafenib in advanced hepatocellular carcinoma. N Engl J Med. 2008 Jul 24;359(4):378-90. doi: 10.1056/NEJMoa0708857. PMID 18650514
- [Background] Cheng AL, Kang YK, Chen Z, Tsao CJ, Qin S, Kim JS, Luo R, Feng J, Ye S, Yang TS, Xu J, Sun Y, Liang H, Liu J, Wang J, Tak WY, Pan H, Burock K, Zou J, Voliotis D, Guan Z. Efficacy and safety of sorafenib in patients in the Asia-Pacific region with advanced hepatocellular carcinoma: a phase III randomised, double-blind, placebo-controlled trial. Lancet Oncol. 2009 Jan;10(1):25-34. doi: 10.1016/S1470-2045(08)70285-7. Epub 2008 Dec 16. PMID 19095497
- [Background] Kudo M, Finn RS, Qin S, Han KH, Ikeda K, Piscaglia F, Baron A, Park JW, Han G, Jassem J, Blanc JF, Vogel A, Komov D, Evans TRJ, Lopez C, Dutcus C, Guo M, Saito K, Kraljevic S, Tamai T, Ren M, Cheng AL. Lenvatinib versus sorafenib in first-line treatment of patients with unresectable hepatocellular carcinoma: a randomised phase 3 non-inferiority trial. Lancet. 2018 Mar 24;391(10126):1163-1173. doi: 10.1016/S0140-6736(18)30207-1. PMID 29433850
- [Background] Choi JH, Chung WJ, Bae SH, Song DS, Song MJ, Kim YS, Yim HJ, Jung YK, Suh SJ, Park JY, Kim DY, Kim SU, Cho SB. Randomized, prospective, comparative study on the effects and safety of sorafenib vs. hepatic arterial infusion chemotherapy in patients with advanced hepatocellular carcinoma with portal vein tumor thrombosis. Cancer Chemother Pharmacol. 2018 Sep;82(3):469-478. doi: 10.1007/s00280-018-3638-0. Epub 2018 Jul 7. PMID 29982870
- [Background] Cheng AL, Guan Z, Chen Z, Tsao CJ, Qin S, Kim JS, Yang TS, Tak WY, Pan H, Yu S, Xu J, Fang F, Zou J, Lentini G, Voliotis D, Kang YK. Efficacy and safety of sorafenib in patients with advanced hepatocellular carcinoma according to baseline status: subset analyses of the phase III Sorafenib Asia-Pacific trial. Eur J Cancer. 2012 Jul;48(10):1452-65. doi: 10.1016/j.ejca.2011.12.006. Epub 2012 Jan 10. PMID 22240282
- [Background] Jeong SW, Jang JY, Shim KY, Lee SH, Kim SG, Cha SW, Kim YS, Cho YD, Kim HS, Kim BS, Kim KH, Kim JH. Practical effect of sorafenib monotherapy on advanced hepatocellular carcinoma and portal vein tumor thrombosis. Gut Liver. 2013 Nov;7(6):696-703. doi: 10.5009/gnl.2013.7.6.696. Epub 2013 Aug 14. PMID 24312711
- [Background] Song DS, Song MJ, Bae SH, Chung WJ, Jang JY, Kim YS, Lee SH, Park JY, Yim HJ, Cho SB, Park SY, Yang JM. A comparative study between sorafenib and hepatic arterial infusion chemotherapy for advanced hepatocellular carcinoma with portal vein tumor thrombosis. J Gastroenterol. 2015 Apr;50(4):445-54. doi: 10.1007/s00535-014-0978-3. Epub 2014 Jul 16. PMID 25027973
- [Background] Lee IC, Chen YT, Chao Y, Huo TI, Li CP, Su CW, Lin HC, Lee FY, Huang YH. Determinants of survival after sorafenib failure in patients with BCLC-C hepatocellular carcinoma in real-world practice. Medicine (Baltimore). 2015 Apr;94(14):e688. doi: 10.1097/MD.0000000000000688. PMID 25860213
- [Background] El-Khoueiry AB, Sangro B, Yau T, Crocenzi TS, Kudo M, Hsu C, Kim TY, Choo SP, Trojan J, Welling TH Rd, Meyer T, Kang YK, Yeo W, Chopra A, Anderson J, Dela Cruz C, Lang L, Neely J, Tang H, Dastani HB, Melero I. Nivolumab in patients with advanced hepatocellular carcinoma (CheckMate 040): an open-label, non-comparative, phase 1/2 dose escalation and expansion trial. Lancet. 2017 Jun 24;389(10088):2492-2502. doi: 10.1016/S0140-6736(17)31046-2. Epub 2017 Apr 20. PMID 28434648
- [Background] Zhu AX, Finn RS, Edeline J, Cattan S, Ogasawara S, Palmer D, Verslype C, Zagonel V, Fartoux L, Vogel A, Sarker D, Verset G, Chan SL, Knox J, Daniele B, Webber AL, Ebbinghaus SW, Ma J, Siegel AB, Cheng AL, Kudo M; KEYNOTE-224 investigators. Pembrolizumab in patients with advanced hepatocellular carcinoma previously treated with sorafenib (KEYNOTE-224): a non-randomised, open-label phase 2 trial. Lancet Oncol. 2018 Jul;19(7):940-952. doi: 10.1016/S1470-2045(18)30351-6. Epub 2018 Jun 3. PMID 29875066
- [Background] Xu J, Zhang Y, Jia R, Yue C, Chang L, Liu R, Zhang G, Zhao C, Zhang Y, Chen C, Wang Y, Yi X, Hu Z, Zou J, Wang Q. Anti-PD-1 Antibody SHR-1210 Combined with Apatinib for Advanced Hepatocellular Carcinoma, Gastric, or Esophagogastric Junction Cancer: An Open-label, Dose Escalation and Expansion Study. Clin Cancer Res. 2019 Jan 15;25(2):515-523. doi: 10.1158/1078-0432.CCR-18-2484. Epub 2018 Oct 22. PMID 30348638
- [Background] Ribas A, Puzanov I, Dummer R, Schadendorf D, Hamid O, Robert C, Hodi FS, Schachter J, Pavlick AC, Lewis KD, Cranmer LD, Blank CU, O'Day SJ, Ascierto PA, Salama AK, Margolin KA, Loquai C, Eigentler TK, Gangadhar TC, Carlino MS, Agarwala SS, Moschos SJ, Sosman JA, Goldinger SM, Shapira-Frommer R, Gonzalez R, Kirkwood JM, Wolchok JD, Eggermont A, Li XN, Zhou W, Zernhelt AM, Lis J, Ebbinghaus S, Kang SP, Daud A. Pembrolizumab versus investigator-choice chemotherapy for ipilimumab-refractory melanoma (KEYNOTE-002): a randomised, controlled, phase 2 trial. Lancet Oncol. 2015 Aug;16(8):908-18. doi: 10.1016/S1470-2045(15)00083-2. Epub 2015 Jun 23. PMID 26115796
- [Background] Robert C, Ribas A, Wolchok JD, Hodi FS, Hamid O, Kefford R, Weber JS, Joshua AM, Hwu WJ, Gangadhar TC, Patnaik A, Dronca R, Zarour H, Joseph RW, Boasberg P, Chmielowski B, Mateus C, Postow MA, Gergich K, Elassaiss-Schaap J, Li XN, Iannone R, Ebbinghaus SW, Kang SP, Daud A. Anti-programmed-death-receptor-1 treatment with pembrolizumab in ipilimumab-refractory advanced melanoma: a randomised dose-comparison cohort of a phase 1 trial. Lancet. 2014 Sep 20;384(9948):1109-17. doi: 10.1016/S0140-6736(14)60958-2. Epub 2014 Jul 15. PMID 25034862
- [Background] Tang B, Yan X, Sheng X, Si L, Cui C, Kong Y, Mao L, Lian B, Bai X, Wang X, Li S, Zhou L, Yu J, Dai J, Wang K, Hu J, Dong L, Song H, Wu H, Feng H, Yao S, Chi Z, Guo J. Safety and clinical activity with an anti-PD-1 antibody JS001 in advanced melanoma or urologic cancer patients. J Hematol Oncol. 2019 Jan 14;12(1):7. doi: 10.1186/s13045-018-0693-2. PMID 30642373
- [Background] Shuqun C, Mengchao W, Han C, Feng S, Jiahe Y, Guanghui D, Wenming C, Peijun W, Yuxiang Z. Tumor thrombus types influence the prognosis of hepatocellular carcinoma with the tumor thrombi in the portal vein. Hepatogastroenterology. 2007 Mar;54(74):499-502. PMID 17523307
- See also: PVTT classification refers to Cheng's classification — http://www.cqvip.com/QK/90800A/20044/9747565.html